CLINICAL TRIAL: NCT02247882
Title: Effectiveness of Health Education Compared to Aquatic Physical Therapy for Patients With Knee Osteoarthritis: a Randomized Clinical Trial
Brief Title: Effectiveness of Aquatic Physical Therapy for Knee Osteoarthritis Patients
Acronym: RCT-OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Collaborators: Ministry of Health, Brazil (Other Government); Fundação Araucária (Other)
Responsible Party: Principal Investigator, Jefferson Rosa Cardoso, Ligia Maria Facci, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RCTOA14; 1406 (Registry Identifier: Ligia Facci)
Record Dates: First submitted 2014-09-21; First posted 2014-09-25 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Patient Education; Aquatic Exercise; kinetic
MeSH Terms: conditions — Osteoarthritis | interventions — Patient Education as Topic; Aquatic Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Education (Experimental): Health Education.
  Interventions: Other: Patient Education
- Aquatic Physical Therapy (Active Comparator): Protocol of aquatic physical therapy exercises.
  Interventions: Other: Aquatic Physical Therapy

INTERVENTIONS:
Other: Patient Education — The educational program will comprise a multidisciplinary team: doctor, pharmacist, nurse, nutritionist, psychologist, physiotherapist and physical educator. Classes will be weekly in groups for eight weeks, with a duration of two hours.
  The education program will include the following items: guidelines about the disease and its complications, strategies for pain management (pharmacological and cognitive), physical exercise, nutrition and weight control, medication (type, interactions, current trends, side effects ), balance, proprioception, fall prevention, coping with chronic pain.
  Other Names: Health Education
  Arms: Patient Education
Other: Aquatic Physical Therapy — The exercise protocol will consist of: five minutes of heating with walking and patellar mobilization; ten minutes stretching the muscles of the lower limbs (quadriceps, gluteus, adductors and abductors of hip sural triceps and hamstrings); ten minutes isometric and dynamic exercises with elastic (quadriceps, gluteus, adductors and abductors of hip sural triceps and hamstrings); twenty minutes away from aerobic exercise (stationary running deep running water); ten minutes in functional training step and proprioceptive exercises; and five minutes of cooling with stretching of muscles of lower limbs (quadriceps, gluteus, adductors and abductors of hip sural triceps and hamstrings).
  Other Names: Aquatic Exercise
  Arms: Aquatic Physical Therapy

SUMMARY:
The purpose of this study is to determine whether education or aquatic physical therapy are effective in the treatment of osteoarthritis in Knee due to intensity of pain, function capacity, quality of life and kinetic.

DETAILED DESCRIPTION:
Sixty patients will be recruited from clinics and through printed newspaper. Physicians who routinely evaluate patients with this diagnosis will be informed of the study, and the same will be announced by television call.

After passing a medical examination confirming the clinical diagnosis of knee osteoarthritis by American College of Rheumatology and other criteria, the elect will be informed of the objectives of the study and invited to participate.

After evaluation of the records of referrals of knee OA, patients receive phone calls, will be informed of the research objectives, questioned regarding the inclusion and exclusion criteria of the study and invited to participate in the study.

Upon study entry, personal information (name, age, gender, address and telephone) will be confirmed by a secretary, who will give the registration number of the patient. Personal information, as well as their radiographs, will be kept in personal form, with number of study enrollment.

Before and after implementation of treatment protocols, as well as after three months, all patients will be assessed by an independent examiner, ie, that have no knowledge about the intervention with respect to different variables. The independent examiner will have been previously trained for this role to become fit to do so.

Individuals will be assessed using the rubric for the outcomes of pain intensity using a Visual Analogue Scale (VAS); functional capacity of the Western Ontario and McMaster Universities Index (WOMAC); balance the Activities-specific Balance Confidence (ABC) and by static posturography and reaction forces to the ground by static force platform. Body weight will be checked by portable scale; height, and waist circumference with tape measure to calculate BMI.

After evaluation, patients will be divided by the numbers generated by the computer through the site (www.random.org) in both treatment groups with 30 patients. After the generation of numbers, they will be transformed into a card with the assigned treatment (1- Patient Education; 2 Aquatic Physiotherapy) and then placed in sealed, opaque, sequentially numbered envelopes. Thus, it prevented the evaluator and the therapist choose the group to which the patient is assigned. Procedures for randomization and allocation, as well as assessments and interventions will be blinded.

The educational program will comprise a multidisciplinary team: doctor, pharmacist, nurse, nutritionist, psychologist, physiotherapist and physical educator. Classes will be weekly in groups for eight weeks, lasting two hours, to be held in the Parlor of Our Lady of Grace Church, belonging to the scope of the Health Unit Vila Brazil.

The program will include education, following the suggestions of Coleman et al. the following items: guidelines about the disease and its complications, strategies for pain management (pharmacological and cognitive), physical exercise, nutrition and weight control, medication (type, interactions, current trends, side effects), balance, proprioception , fall prevention, coping with chronic pain. Following, practical activities on the themes will be addressed.

To enhance the information at the end, patients will receive printed material with the guidelines given by the professional. Still, the first and last day of the education program, patients will respond a questionnaire addressing their knowledge about the disease developed by the researchers.

Supervised aquatic exercise will run individually, twice a week, lasting 60 minutes, for eight weeks, totaling 16 sessions at the Center for Aquatic Physical Therapy Professor Paulo Armindo Seibert, Universidade Estadual de Londrina. The water temperature will be maintained at approximately 32 degrees, with a depth of 1.20m. The exercise protocol will consist of: five minutes of heating with walking and patellar mobilization; ten minutes stretching the muscles of the lower limbs (quadriceps, gluteus, adductors and abductors of hip sural triceps and hamstrings); ten minutes isometric and dynamic exercises with elastic (quadriceps, gluteus, adductors and abductors of hip sural triceps and hamstrings); twenty minutes away from aerobic exercise (stationary running deep water running); ten minutes in functional training step and proprioceptive exercises; and five minutes of cooling with stretching of muscles of lower limbs (quadriceps, gluteus, adductors and abductors of hip sural triceps and hamstrings).

Both groups will receive guidance home exercises two to three times a week, and reinforced by familiar previously illustrated booklets, which include the same goals of aquatic exercises: heating, self stretching of the lower limb muscles, isometric and dynamic exercises of the lower limbs , proprioceptive and functional exercises, aerobic exercises is relaxation.

Three months after the end of intervention protocols, ie, at the end of follow-up, patients in the group Education will be invited to perform aquatic therapy and patients in group aquatic therapy will receive the manual of educational guidelines.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 60 and 85 years;
* patients with knee OA by a physician confirmed by the criteria of American College of Rheumatology;
* patients with clinical and cognitive activities for the realization of the pool conditions, confirmed by the Mini-Exam Mental state.

Exclusion Criteria:

* patients undergoing surgical procedures in the last six months;
* patients with chronic diseases such as coronary, other rheumatic diseases such as rheumatoid arthritis; serious diseases such as cancer; chronic obstructive pulmonary diseases; uncontrolled hypertensive;
* patients unable to walk without aid equipment;
* patients who have contraindications to practice exercises;
* patients who have contraindications for entry into the pool, such as urinary or fecal incontinence and skin problems;
* patients participating in nutrition programs or physical activity in the last two months (or resisted aerobic activity more than once a week for at least two months);
* patients with metal implants in the lower limbs;
* patients with morbid obesity (body mass index (BMI)> 40 kg / m 2);
* Patients unable to continue the study by programmed change of address or hospitalization.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pain | up to 3 months
  Evaluation of pain - EVA

SECONDARY OUTCOMES:
Function | 2 and 3 months
  Physical Function - WOMAC Index
Balance | 2 and 3 months
  ABC Scale and postural balance
Quality Of Live | 2 and 3 months
  SF-36 Questionaire
kinetic | 2 and 3 months
  Ground Reaction Forces and postural balance

CONTACTS AND LOCATIONS:
Overall Officials: Ligia M Facci, PT, PhD, Principal Investigator — Adjunct Professor
Locations (1):
- Aquatic Physical Therapy Center "Paulo A. Seibert", Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Lyytinen T, Liikavainio T, Bragge T, Hakkarainen M, Karjalainen PA, Arokoski JP. Postural control and thigh muscle activity in men with knee osteoarthritis. J Electromyogr Kinesiol. 2010 Dec;20(6):1066-74. doi: 10.1016/j.jelekin.2010.05.005. Epub 2010 Jun 11. PMID 20541439
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Fernandes MI. Tradução e validação do questionário de qualidade de vida específico para osteoartrose WOMAC (Western Ontario McMasterUniversities) para a língua portuguesa. São Paulo, 2002. 103p. Tese de Mestrado - Universidade Federal de São Paulo - Escola Paulista de Medicina - Reumatologia.
- [Background] Marques AP, Mendes YC, Taddei U, Pereira CA, Assumpcao A. Brazilian-Portuguese translation and cross cultural adaptation of the activities-specific balance confidence (ABC) scale. Braz J Phys Ther. 2013 Mar-Apr;17(2):170-8. doi: 10.1590/S1413-35552012005000072. PMID 23778771
- [Background] Duarte M, Freitas SMSF. Revisão sobre posturografia baseada em plataforma de força para avaliação do equilíbrio. Rev Bras Fisioter, São Carlos, v. 14, n. 3, p. 183-92, maio/jun. 2010.
- [Background] CICONELLI RM, FERRAZ MB, SANTOS W, MEINÃO I, QUARESMA MR. Tradução para a língua portuguesa e validação do questionário genérico de avaliação da qualidade de vida SF-36 (Brasil SF-36).RevBrasreumatol 1999; 39(3): 143-150.